CLINICAL TRIAL: NCT07353151
Title: Artificial Intelligence-based, Virtual Reality Application to Provide Data- Driven, Patient-centred Treatment for People With Eating Disorders
Acronym: OASIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRAS: 359405
Record Dates: First submitted 2025-11-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Anorexia Nervosa; Feeding and Eating Disorders
Keywords: Anorexia nervosa (AN); Virtual reality (VR); Eating disorders; Food exposure; Feasibility study; Food-related anxiety; Exposure-based intervention; South London and Maudsley (SLaM); King's College London (KCL); United Kingdom
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Single-group, open-label feasibility design. All participants receive the OASIS VR add-on alongside treatment as usual across inpatient, day service, or outpatient settings. The intervention consists of five supervised sessions over one week (≈20-30 minutes each). No randomization or control arm in this phase; focus is on feasibility, acceptability, adherence, and safety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OASIS VR + Treatment as Usual (TAU) (Experimental): Single-group, open-label feasibility arm. Participants receive a brief virtual reality (VR) program (OASIS) alongside treatment as usual. The VR program is delivered as five supervised sessions over one week (≈20-30 minutes per session) in inpatient, day service, or outpatient settings.
  Interventions: Behavioral: OASIS virtual reality (VR) program

INTERVENTIONS:
Behavioral: OASIS virtual reality (VR) program — Immersive VR sessions including (a) food-related exposure scenes, (b) relaxing music, and (c) motivational prompts and goal-setting. Delivered once daily on weekdays for one week (five sessions; ≈20-30 minutes each), supervised by a clinician or trained researcher. Sessions may be paused or stopped at any time.

SUMMARY:
The goal of this clinical trial is to see if a short virtual reality (VR) program can be used safely and comfortably with people receiving care for anorexia nervosa. The study will also check if people are willing to take part and complete the full week of VR sessions.

The main questions the study will answer are:

Can the investigators recruit and keep participants in the study? Do participants complete most of the VR sessions? Do they find the experience helpful and acceptable? Are there any side effects, like nausea or dizziness?

Participants will:

* Take part in one VR session each weekday (about 20 to 30 minutes) for one week
* Continue their usual care during this time
* Answer questions before and after the VR sessions about their anxiety, mood, motivation, and experience
* Some participants may join a short interview or focus group to share feedback

The VR program includes scenes for food-related exposure, calming music, motivational phrases, and goal setting. The app was designed with help from people with lived experience of anorexia and based on psychological therapies used in treatment.

Who can take part:

* Adults aged 18 or older
* People receiving or waiting for care for anorexia nervosa at South London and Maudsley NHS Foundation Trust (SLaM)
* People who are medically stable and able to give informed consent

Why this matters:

This study will help researchers understand if using VR in eating disorder services is practical, safe, and acceptable. The results will help plan a larger trial in the future to see if this type of VR treatment can support recovery from anorexia nervosa. Taking part is voluntary, and participants can stop at any time.

DETAILED DESCRIPTION:
This single-site, open-label feasibility clinical trial will test a brief virtual reality (VR) program (OASIS) delivered alongside treatment as usual for adults with anorexia nervosa. OASIS was co-developed by South London and Maudsley NHS Foundation Trust (SLaM), King's College London, and SyncVR Medical UK with input from people with lived experience.

The VR sessions are designed to support recovery by providing:

* Food-related exposure scenes to practise approaching commonly avoided foods
* Relaxing environments with music
* Motivational prompts and goal-setting within the VR experience

Participants complete five supervised VR sessions over one week (about 20-30 minutes each) in inpatient, day service, or outpatient settings. A clinician or trained researcher is present for all sessions. Pacing can be adjusted, and sessions can be paused or stopped at any time.

Feasibility will be assessed using study process measures (for example, recruitment and retention, session completion, and brief usability/acceptability feedback) and session logs. Safety is monitored during every session and via routine clinical information already collected in care; no additional research blood tests are required.

Participants complete brief assessments at baseline and after the one-week intervention. These include validated self-report measures of eating-disorder symptoms, food-related fear, mood/anxiety, and motivation, plus very short ratings around sessions to track immediate experience (for example, anxiety or relaxation). A subset may take part in a short interview or focus group to describe what felt helpful or difficult and suggest refinements.

There is no randomization or control arm in this feasibility phase. Findings will be used to decide whether and how to run a larger randomized controlled trial, including practical procedures (for example, session dose and outcome burden), expected adherence, safety monitoring steps, and willingness to be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years.
* Anorexia nervosa receiving or awaiting treatment as usual (TAU) within South London and Maudsley NHS Foundation Trust (inpatient, day service, or outpatient).
* Medically stable and clinically suitable to take part in brief VR sessions alongside TAU (as judged by the treating team).
* Able to give informed consent.

Exclusion Criteria:

* Current or recent (within 12 months) serious self-harm with suicidal intent, or behaviour that posed a risk to life (e.g., overdose, deep cutting, swallowing sharp objects), or self-harm likely to cause lasting impairment.
* Active suicidality or high risk of suicide.
* Untreated or unstable epilepsy.
* Psychotic disorder.
* Outpatient participants with BMI < 10.
* Current participation in another research study or clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Session adherence to the VR intervention | Baseline to end of Week 1 (5 weekdays)
  Proportion of scheduled VR sessions completed per participant, recorded from session logs. A session counts as completed if ≥20 minutes are delivered. Primary endpoint = % of participants who complete ≥4 of 5 sessions; the investigators will also report mean (SD) sessions completed.

SECONDARY OUTCOMES:
Recruitment and retention feasibility | Months 2-10 (recruitment) and Baseline to end of Week 1 (retention)
  Recruitment = % of eligible approached who consent. Retention = % of consented who complete the 1-week assessment.
EDE-Q Global Score | Baseline and end of Week 1
  Change in global score on the Eating Disorder Examination Questionnaire (EDE-Q) from baseline to end of Week 1. Score (0-6); higher scores indicate greater severity of eating disorder symptoms.
EFQ Total Score | Baseline and end of Week 1
  Change in total score on the Eating and Food Questionnaire (EFQ) from baseline to end of Week 1.
  Units: Score (0-50); higher scores indicate more maladaptive eating behaviors.
FOFM Score | Baseline and end of Week 1
  Change in score on the Fear of Food Measure (FOFM) from baseline to end of Week 1.
  Units: Score (0-40); higher scores indicate greater food-related anxiety.
M3VAS Items | Baseline and end of Week 1
  Change in visual analog scale ratings (M3VAS) for mood and anxiety from baseline to end of Week 1.
  Units: Score (0-100 mm); higher scores indicate greater symptom severity.
DASS-42 Total Score | Baseline and end of Week 1
  Change in total score on the Depression Anxiety Stress Scales (DASS-42) from baseline to end of Week 1. Units: Score (0-126); higher scores indicate greater psychological distress.
Acceptability/usability of VR | End of Week 1
  Study-specific 0-10 ratings of acceptability/helpfulness (higher = better); summarized as mean (SD).
Willingness outcomes | End of Week 1
  (a) Willingness to try foods encountered in VR outside sessions (four 0-10 items: willingness, readiness, confidence, 1-week likelihood); (b) willingness to participate in a future randomized trial (Yes/No).
Feasibility of assessment battery | Baseline and end of Week 1
  Completion rates across all planned questionnaires; instruments with >25% missing at either time point flagged as infeasible for a future trial.
Safety (adverse events and VR-related symptoms) | During sessions through end of Week 1
  Counts/types of adverse events (including nausea, dizziness, headache); % of participants with ≥1 event.
Body Mass Index (BMI) | Baseline and end of Week 1
  Change in body mass index (BMI) from baseline to end of Week 1. Units: kg/m²; higher values indicate higher body mass.

CONTACTS AND LOCATIONS:
Overall Officials: Hubertus Himmerich, MD, PhD, Principal Investigator — South London and Maudsley NHS Foundation Trust; King's College London; Janet Treasure, MD, PhD, Study Chair — South London and Maudsley NHS Foundation Trust; King's College London

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of de-identified individual participant data (IPD) is under consideration pending sponsor and NHS approvals, information governance review, and repository selection. Aggregate results will be published. An IPD sharing statement will be updated once approvals are in place.

REFERENCES:
- [Background] Cardi V, Krug I, Perpina C, Mataix-Cols D, Roncero M, Treasure J. The use of a nonimmersive virtual reality programme in anorexia nervosa: a single case-report. Eur Eat Disord Rev. 2012 May;20(3):240-5. doi: 10.1002/erv.1155. Epub 2011 Sep 20. PMID 21932282
- [Background] Bektas S, Natali L, Rowlands K, Valmaggia L, Di Pietro J, Mutwalli H, Himmerich H, Treasure J, Cardi V. Exploring Correlations of Food-Specific Disgust with Eating Disorder Psychopathology and Food Interaction: A Preliminary Study Using Virtual Reality. Nutrients. 2023 Oct 19;15(20):4443. doi: 10.3390/nu15204443. PMID 37892518
- [Background] Natali L, Meregalli V, Rowlands K, Di Pietro J, Treasure J, Collantoni E, Meneguzzo P, Tenconi E, Favaro A, Fontana F, Ceccato E, Sala A, Valmaggia L, Cardi V. Virtual food exposure with positive mood induction or social support to reduce food anxiety in anorexia nervosa: A feasibility study. Int J Eat Disord. 2024 Mar;57(3):703-715. doi: 10.1002/eat.24155. Epub 2024 Feb 17. PMID 38366755
- [Background] Young KS, Rennalls SJ, Leppanen J, Mataix-Cols D, Simmons A, Suda M, Campbell IC, O'Daly O, Cardi V. Exposure to food in anorexia nervosa and brain correlates of food-related anxiety: findings from a pilot study. J Affect Disord. 2020 Sep 1;274:1068-1075. doi: 10.1016/j.jad.2020.05.077. Epub 2020 May 25. PMID 32663934
- See also: South London & Maudsley NHS Foundation Trust - Adult Eating Disorders Service — https://www.slam.nhs.uk/
- See also: King's College London - Eating & Weight Research (CREW) — https://www.kcl.ac.uk/